CLINICAL TRIAL: NCT02329626
Title: Evaluation Via PET Scan of Metabolic Anomolies Associated With the 6 Month Clinical Evolution of Patients Suffering From Motor Conversion Disorder
Brief Title: Metabolic Anomolies Associated With the 6 Month Clinical Evolution of Patients Suffering From Motor Conversion Disorder
Acronym: HYCORE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2014/ETIC-01; 2014-A01159-38 (Other: ANSM)
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2018-03

CONDITIONS: Conversion Disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken at baseline, 3 months and 6 months.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: The study population consists of patients with paralysis, motor weakness or abnormal movements meeting DSM-IV criteria for motor conversion disorder consulting via the Emergency or Neurology department of participating centers.
  Intervention: PET CT 18 FDG
  Interventions: Device: PET CT 18 FDG

INTERVENTIONS:
Device: PET CT 18 FDG — Positron emission tomography with 2-deoxy-2-[fluorine-18]fluoro- D-glucose integrated with computed tomography.
  This intervention is required for the observational needs of the study.

SUMMARY:
The main objective of this study is to make a first evaluation of the relationship between metabolic abnormalities objectified by Positron emission tomography with 2-deoxy-2-[fluorine-18]fluoro- D-glucose integrated with computed tomography (PET CT 18 FDH) performed at rest at the onset of symptoms in patients with a first episode of motor conversion disorder and the persistence of a motor disability at 6 months measured by the modified Rankin score (mRS).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To assess whether metabolic abnormalities objectified by PET CT 18 FDH performed at rest at the onset of symptoms may be predictive of persistent disability at 6 months as measured by the EDSS, the NIHSS and WHO status.

B. To assess whether metabolic abnormalities objectified by PET CT 18 FDH performed at rest at 3 months after diagnosis may be predictive of persistent motor disability at 6 months (EDSS, NIHSS, mRS, WHO) C. To search for and characterize any abnormalities of metabolism objectified in the initial PET CT 18 FDH predictive of persistent motor disability at 3 months.

D. To determine if there are persistent metabolic abnormalities 3 months post-diagnosis independently of the clinical course (marker trait).

E. Define the brain areas whose metabolism is often altered in patients with motor conversion disorders.

F. Establish a collection of biological samples from patients for future research studies of prognostic biomarkers of a motor conversion disorder.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given free and informed consent and signed the consent
* The patient must be affiliated with or beneficiary of a health insurance plan
* The patient meets DSM-IV criteria for motor conversion disorder (with paralysis, motor weakness or abnormal movements) lasting for less than 1 month and euthymic (HAMD score < or = 7, as evaluated by a psychiatrist)
* First episode (incident cases)
* The latest symptom dates to within a month
* The patient is not under neuroleptics

Exclusion Criteria:

* The subject is participating in another study
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection, guardianship or curatorship
* The subject refuses to sign the consent
* It is not possible to correctly inform the patient
* The patient is pregnant, parturient or she is breastfeeding
* Specialized clinical neurological examination and brain and spinal cord MRI revealed an organic neurological cause
* The subject has a HAMD score > 7
* The subject currently has manic/hypomanic episode, a diagnosis of substance abuse or dependency (excluding tobacco), a diagnosis of schizophrenia (any time in the past) or chronic neurological disease (active epilepsy, stroke, brain tumor)
* Suicidal or high risk for suicide (according to MINI assessment)
* Contra-indication for a PET scan
* Patient under neuroleptics at inclusion
* The last symptom happened over 1 month ago
* The patient has had previous episodes (prevalent cases)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with paralysis, motor weakness or abnormal movements meeting DSM-IV criteria for motor conversion disorder consulting via the Emergency or Neurology department of participating centers.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Presence/absence of a modified Ranking score > 1 | 6 months
Presence/absence of a metabolic anomoly according to PET CT 18 FDG | Day 0 to Day 15
  PET CT 18 FDG = Positron emission tomography with 2-deoxy-2-[fluorine-18]fluoro- D-glucose integrated with computed tomography

SECONDARY OUTCOMES:
Presence/absence of a metabolic anomoly according to PET CT 18 FDG | 3 months
Modified Rankin Score | 3 months
Modified Rankin Score | 6 months
EDSS score | Day 0 to Day 15
EDSS score | 3 months
EDSS score | 6 months
NIHSS score | Day 0 to Day 15
NIHSS score | 3 months
NIHSS score | 6 months
MINI questionnaire | Day 0 to Day 15
HAMD scale | Day 0 to Day 15
HAMD scale | 3 months
HAMD scale | 6 months
HADS scale | Day 0 to Day 15
HADS scale | 3 months
HADS scale | 6 months
WHO score | 3 months
WHO score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ismaël Conejero, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CHRU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Conejero I, Thouvenot E, Abbar M, Mouchabac S, Courtet P, Olie E. Neuroanatomy of conversion disorder: towards a network approach. Rev Neurosci. 2018 Jun 27;29(4):355-368. doi: 10.1515/revneuro-2017-0041. PMID 29252202